CLINICAL TRIAL: NCT06607107
Title: A Single-arm Phase II Clinical Study Evaluating the Efficacy and Safety of Systemic Chemotherapy(mFOLFOX7) Combined With Camrelizumab and Apatinib in BCLC Stage A/B Hepatocellular Carcinoma Patients Beyond Milan Criteria
Brief Title: mFOLFOX7 Plus Camrelizumab and Apatinib in BCLC Stage A/B Hepatocellular Carcinoma Patients Beyond Milan Criteria
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Jiangsu Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2024-107-01
Record Dates: First submitted 2024-09-11; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Hepatocellular Carcinoma Non-resectable
MeSH Terms: interventions — camrelizumab; apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mFOLFOX7 combined with Apatinib and Camrelizumab (Experimental): mFOLFOX7(Oxaliplatin, Calcium Levofolinate, Fluorouracil) combined with Apatinib and Camrelizumab
  Interventions: Drug: mFOLFOX7 combined with Camrelizumab and apatinib

INTERVENTIONS:
Drug: mFOLFOX7 combined with Camrelizumab and apatinib — mFOLFOX7(Oxaliplatin 85mg/m2, Calcium Levofolinate 200mg/m2, Fluorouracil 400 mg/m2 D1，2400mg/m2 maintain 46 hours，) combined with Apatinib and Camrelizumab 200mg every 3 weeks. Taking Apatinib-Mesylate Tablets (250 mg/tablet) orally after meals, once a day, for continuous medication.
  Other Names: mFOLFOX7 plus Camrelizumab and apatinib

SUMMARY:
This study was designed to evaluate the effectiveness and safety of mFOLFOX7（Oxaliplatin,Calcium Levofolinate,Fluorouracil） combined with Apatinib and Camrelizumab for Hepatocellular Carcinoma.

The primary outcome measure is to evaluate the primary pathological response (MPR) rate of the therapy for Hepatocellular Carcinoma.

The secondary Outcome measures include the objective response rate (ORR), the duration of response (DOR), disease control rate (DCR), progression-free survival rate (PFSR) [ Time Frame: 6- and 12-month], overall survival rate (OSR) [ Time Frame: 6- and 12-month], the median progression-free survival time (mPFS) and median overall survival time (mOS) of the therapy for Hepatocellular Carcinoma.

Moreover, this study aims to assess the safety and tolerability of the Therapy for Hepatocellular Carcinoma.

DETAILED DESCRIPTION:
Hepatocellular carcinoma(HCC) is a common high-grade malignant tumor in my country, with limited treatment options and poor prognosis.

Early and middle stage (BCLC A or B) surgical resection is the main curative method for liver cancer, except for a few very early stages. Small liver cancer has a high short-term recurrence rate after surgery, with a median survival time of about 2 years and a 5-year survival rate of<20%. Treatment objectives for advanced liver cancer.

Previously, systemic therapy and transcatheter arterial chemoembolization(TACE) were mainly used for treatment, while targeted therapy and immunotherapy in systemic therapy have made rapid progress in recent years.

Trastuzumab and chemotherapy can increase the ORR of human epidermal growth factor receptor 2(HER2) positive advanced gastric cancer from 51.9% to 74.4%.

Preliminary small sample studies have shown that veins the combination of mFOLFOX7 regimen with Carolizumab and Apatinib may be a potential treatment for CNLC stage III hepatocellular carcinoma.A strategy that is effective, safe, and easy to implement, with preliminary research results similar to FOLFOX-HAIC combined with targeted immunotherapy. Especially for patients with concomitant main portal vein tumor thrombus showed very good results, and the extremely low microvascular invasion(MVI) in postoperative pathology also suggests the possibility of good therapeutic value for microvascular metastasis of liver cancer.

The Milan standard is an international standard used in liver transplantation, and patients who meet the standard have a lower recurrence rate and a longer lifespan.Survival period, specifically as follows: (1) The diameter of a single tumor does not exceed 5 cm; (2) The number of multiple tumors should not exceed 3 and the most Large diameter not exceeding 3cm; (3) The tumor has no invasion of large hepatic vessels or distant metastasis. We can also find that the Milan standard can significantly distinguish the treatment effect of liver cancer, and surpassing Milan's standard liver cancer has a significantly higher early recovery rate. There are also studies showing that liver cancer patients who exceed Milan's standards are receiving downgraded treatment of the overall survival rate and disease progression free survival rate after liver transplantation in patients who meet Milan's criteria are correlated with the overall survival rate after liver transplantation nearly. Therefore, in our study, neoadjuvant therapy targeting liver cancer with a high risk of recurrence has a high clinical value. The significance and expectation of camrelizumab and apatinib combined with intravenous mFOLFOX7 chemotherapy regimen are to improve the MPR rate of liver cancer treatment and reduce patient risk.

The MVI rate is increased to achieve a phase reduction effect and prolong the patient's life

ELIGIBILITY:
Inclusion Criteria:

1. Before treatment, histologically or cytologically or clinically diagnosed as hepatocellular carcinoma (HCC) and the clinical stage belongs to BCLC stage A/B HCC that exceeds the Milan criteria.
2. Child-pugh liver function grading: Grade A or B
3. Did not received any type of other first-line drugs such as Sorafenib or Lenvatinib.
4. According to RECIST 1.1 standard and mRECIST standard, patients have at least one measurable lesion (CT scan long diameter ≥10mm and the lesion has not received radiotherapy, freezing or other local treatments)；
5. ECOG PS score 0-2;
6. Expected survival ≥ 12 weeks;
7. Blood routine:White blood cells count ≥3.0×10^9/L Platelet count ≥70×10^9/L Hemoglobin ≥80g/L(without blood transfusion within 14 days); kidney function: Serum creatinine (SCr) ≤ 1.5 times upper limit of normal value (ULN); Liver function:Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal value (ULN); AST or ALT levels ≤ 3 times the upper limit of normal value (ULN)
8. Patients with hepatitis B or C coinfection need to use antiviral drugs and have not used interferon.
9. Women of childbearing age should have a negative serum or urine pregnancy test within 7 days before enrollment and they must be non-lactating patients and agree to use contraceptive measures during the study period and within 6 months after the end of the study. Men should agree to use contraceptive measures during the study period and within 6 months after the end of the study period.
10. Patients volunteered to participate in this study and signed informed consent;

Exclusion Criteria:

1. Have received immunotherapeutic drugs or interferon in the past.
2. Allergic to the drugs in the treatment ;
3. Female subjects with pregnancy or on feeding.
4. Have received other immunotherapy drugs (targeting PD1/PDL1).
5. Patients with combined uncontrolled cardiac clinical symptoms or diseases, such as: (1) heart failure above NYHA class II; (2) unstable angina pectoris; (3) myocardial infarction within 1 year; (4) patients with clinically significant supraventricular or ventricular arrhythmias requiring clinical intervention; (5) those with poorly controlled hypertension by drugs and assessed by doctors as having a high risk of using apatinib.
6. Past medical history includes other tumors or a second tumor, except for cured basal cell carcinoma of the skin, cervical carcinoma in situ and papillary thyroid cancer.
7. Combined with severe infection (CTCAE greater than grade 2) before the start of treatment, such as severe pneumonia requiring hospitalization, active tuberculosis, bacteremia, infectious complications, etc.; baseline chest imaging examination indicates active pulmonary inflammation. There are symptoms and signs of infection within 2 weeks before the first use of the study drug or oral or intravenous antibiotic treatment is required (excluding prophylactic use of antibiotics).
8. Have a history of immunodeficiency, such as positive HIV monitoring, have other acquired or congenital immunodeficiency diseases (such as interstitial pneumonia, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to these diseases and syndromes), or have a history of organ transplantation or bone marrow transplantation; or are taking hormones or other immunosuppressive drugs orally or intravenously; but excluding vitiligo or cured childhood asthma/allergies, and patients who do not require any intervention as adults.
9. Severe coagulation disorders (INR>2.0, PT>16s), those with obvious bleeding tendencies (including but not limited to vomiting blood and having bloody stools every day in the past 3 months).
10. Have the history of abusing psychotropic drugs and unable to quit ,or with mental disorders; with brain metastases or hepatic encephalopathy.
11. As judged by the investigator, the patient may have other factors that may cause the study to be terminated prematurely, such as other serious diseases or serious abnormal laboratory tests or accompanied by other family or social factors that will affect the safety of the subject or the collection of trial data and samples.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2024-02-17 (Actual); Primary Completion 2026-01-11 (Estimated); Study Completion 2028-01-11 (Estimated)

PRIMARY OUTCOMES:
Major pathological response (MPR) rate | 6 months
  MPR rate is defined as the proportion of participants with =<10% residual viable tumor in the tumor bed at the time of surgery, as assessed by central pathological review.

SECONDARY OUTCOMES:
Objective Response Rate(ORR) by RECIST 1.1 | 6 months
  ORR is the proportion of patients who achieved a complete or partial response during or after treatment
pathologic complete response (pCR) rate | 6 months
  pCR is the proportion of surgical specimens with no tumor lesion or only carcinoma in situ.
Duration of remission(DOR) by mRECIST | 12 months
  DOR is the time between the first assessment of the tumor as a complete or partial response and the first assessment as tumor progression or death.
Disease Control Rate(DCR) by mRECIST | 6 months
  DCR is the proportion of all patients who have tumors that shrink or remain stable and stay that way for a certain period of time.
Disease-free-survival(DFS) by RECIST 1.1 | 12 months
  DFS is the time from the beginning of radical surgery to the first recurrence of the tumor and metastasis or death of patient for any reason.
Progression-Free Survival (PFS) by RECIST 1.1 | 12 months
  PFS is intended to be the time during or after treatment when there is no disease progression.
Overall Survival (OS) by RECIST 1.1 | 24 months
  OS is from the point at which treatment begins or the disease is diagnosed to the time at which the patient dies.
Progression-Free Survival rate (PFSR) by RECIST 1.1 | 12 months
  PFSR is the proportion of progression-free survival patients.
Overall Survival Rate (OSR) by RECIST 1.1 | 24 months
  OSR is the proportion of all surviving patients.

CONTACTS AND LOCATIONS:
Overall Officials: linhui Peng, Prof, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No